CLINICAL TRIAL: NCT04263558
Title: Echo: Optimizing a Group-based School Intervention for Children With Emotional Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionsenter for barn og unges psykiske helse (Other)
Collaborators: University of Tromso (Other); Technical University of Trondheim (Unknown)
Responsible Party: Principal Investigator, Simon-Peter Neumer, Dr. Phil., Regionsenter for barn og unges psykiske helse
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 31/18
Record Dates: First submitted 2019-11-27; First posted 2020-02-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Anxiety Depression

STUDY DESIGN:
Intervention Model Description: The study will have a stratified, randomized cluster design. The schools are clusters randomized to different experimental conditions. The factors are (1) feedback from a MFS-system, yes/no, (2) Evidence Based Intervention, long/short (EBI), and (3) parental involvement, high/low. The three factors are related components that, together, should form the strongest intervention outcomes. Each of the 40 recruited schools will therefore be randomly assigned to one of eight experimental conditions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- LHF (Active Comparator): Long intervention (16 sessions) High parental involvement (5 sessions) Feedback
  Interventions: Behavioral: Emotion child
- LHN (Active Comparator): Long intervention (16 sessions) High parental involvement (5 sessions)
  Interventions: Behavioral: Emotion child
- LLF (Active Comparator): Long intervention (16 sessions) Low parental involvement (Brochure) Feedback
  Interventions: Behavioral: Emotion child
- LLN (Active Comparator): Long intervention (16 sessions) Low parental involvement (Brochure)
  Interventions: Behavioral: Emotion child
- SHF (Active Comparator): Short intervention (8 sessions, group) and 8 sessions web-based High parental involvement (5 sessions) Feedback
  Interventions: Behavioral: Emotion child
- SHN (Active Comparator): Short intervention (8 sessions, group) and 8 sessions web-based High parental involvement (5 sessions)
  Interventions: Behavioral: Emotion child
- SLF (Active Comparator): Short intervention (8 sessions, group) and 8 sessions web-based Low parental involvement (Brochure) Feedback
  Interventions: Behavioral: Emotion child
- SLN (Active Comparator): Short intervention (8 sessions, group) and 8 sessions web-based Low parental involvement (Brochure)
  Interventions: Behavioral: Emotion child

INTERVENTIONS:
Behavioral: Emotion child — The MFS will include an idiographic measure of personal aims, symptom burden, displayed on a visual data dashboard to guide further intervention. The EMOTION intervention for children 9 to 12 years with symptoms of anxiety and/or depression will be used in a standard/long version (16 sessions) and a short (8 sessions) but optimized version, using a partial web-based solution with virtual reality (VR)-technology for behavioral experiments and exposure (in short and long version). Parental involvement: Parental participation in a 5-session parent group (high involvement) versus sharing information with parents via a brochure (low Parental involvement).
  Other Names: Measurement Feedback System (MFS); Emotion parent

SUMMARY:
The present study (Echo) will promote much needed research and innovation that optimize service provision in first line health services for the alarmingly high number of school children who suffer from clinical and subthreshold levels of anxiety and depression. The effect of different versions of an evidence-based intervention for this group of children will be tested using a cluster randomized design involving 40 schools across Norway. The aim is to create a framework that allows more evidence-based psychosocial interventions to be provided at a lower cost to society. Echo will provide knowledge about three main evidence gaps for children: (1) The effect of school-based preventive interventions on anxiety and depression; (2) The effect of feedback informed systems, and; (3) the effect and cost-effectiveness of digital health interventions using online sessions and virtual reality technology.

ELIGIBILITY:
Inclusion Criteria:

• Children scoring one standard deviation or more above population mean using established measures for anxiety and/or depression

Exclusion Criteria:

* Retardation or language problems
* Developmental conditions
* Individual considerations approved by the local PI

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1364 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Multidimensional Anxiety Scale | Time 1 baseline
  Anxiety symptoms, minimum 0 to maximum 117, high score indicates worse outcome
Multidimensional Anxiety Scale | Time 2 after approximal 10 weeks
  Anxiety symptoms, minimum 0 to maximum 117, high score indicates worse outcome
Multidimensional Anxiety Scale | Time 3 after approximal 1 year
  Anxiety symptoms, minimum 0 to maximum 117, high score indicates worse outcome
Mood and Feeling Questionnaire | Time 1 baseline
  Depression symptoms, minimum 0 to maximum 26, high score indicates worse outcome
Mood and Feeling Questionnaire | Time 2 after approximal 10 weeks
  Depression symptoms, minimum 0 to maximum 26, high score indicates worse outcome
Mood and Feeling Questionnaire | Time 3 after approximal one year
  Depression symptoms, minimum 0 to maximum 26, high score indicates worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simon-Peter Neumer, Phd, Principal Investigator — Center for Child and Adolescent Mental Health
Locations (3):
- Norway (3):
  - Regionsenter for barn og unges psykiske helse, Oslo
  - Regional kunnskapssenter for barn og unge - Nord, Tromsø
  - Regional kunnskapssenter for barn og unge - Midt, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinsen KD, Aas E, Ingul JM, Lisoy C, Adolfsen F, Rasmussen LM, Wentzel-Larsen T, Neumer SP. Cost-effectiveness analysis of preventive strategies for child anxiety and depression: a health service perspective. Child Adolesc Psychiatry Ment Health. 2025 Oct 1;19(1):107. doi: 10.1186/s13034-025-00962-w. PMID 41034930
- [Derived] Ytreland K, Bania EV, Lydersen S, Sund AM, Neumer SP, Adolfsen F, Martinsen KD, Rasmussen LP, Ingul JM. Parental Involvement in Child Anxiety and Depression: Exploring the Impact of Delivery Format on Modifiable Parental Factors. Child Psychiatry Hum Dev. 2025 Feb 13. doi: 10.1007/s10578-025-01814-6. Online ahead of print. PMID 39946004
- [Derived] Haug IM, Neumer SP, Handegard BH, Lisoy C, Rasmussen LP, Bania EV, Adolfsen F, Patras J. Dose-Response Effects of MittEcho, a Measurement Feedback System, in an Indicated Mental Health Intervention for Children in Municipal and School Services in Norway. Adm Policy Ment Health. 2025 Jan;52(1):223-240. doi: 10.1007/s10488-024-01389-9. Epub 2024 May 29. PMID 38809322
- [Derived] Lisoy C, Neumer SP, Adolfsen F, Ingul JM, Potulski Rasmussen LM, Wentzel-Larsen T, Patras J, Sund AM, Ytreland K, Waaktaar T, Holen S, Askeland AL, Haug IM, Bania EV, Martinsen K. Optimizing indicated cognitive behavioral therapy to prevent child anxiety and depression: A cluster-randomized factorial trial. Behav Res Ther. 2024 May;176:104520. doi: 10.1016/j.brat.2024.104520. Epub 2024 Mar 18. PMID 38522127
- [Derived] Martinsen K, Lisoy C, Wentzel-Larsen T, Neumer SP, Rasmussen LP, Adolfsen F, Sund AM, Ingul JM. School children's mental health during the COVID-19 pandemic. Front Psychol. 2024 Jan 5;14:1290358. doi: 10.3389/fpsyg.2023.1290358. eCollection 2023. PMID 38327509